CLINICAL TRIAL: NCT03957954
Title: Safety and Feasibility of Cultivated Autologous Limbal Stem Cells (cLSC) for Limbal Stem Cell Deficiency
Brief Title: Stem Cell Therapy for Limbal Stem Cell Deficiency
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Eye Institute (NEI) (NIH); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Sophie Deng, MD, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V001; R01EY021797 (NIH)
Record Dates: First submitted 2019-02-21; First posted 2019-05-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Limbal Stem-cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cultivated Limbal Stem-Cells (cLSC) (Experimental): One dose of cultivated limbal stem-cells (cLSC), size between 7.6 to 15 mm in the average diameter.
  Interventions: Biological: cLSC
- Scleral Contact Lens Device (SCL) (Active Comparator): Scleral contact lens device (SCL) will be fitted to stabilize and improve ocular surface.
  Interventions: Device: Scleral contact lens (SCL)

INTERVENTIONS:
Biological: cLSC — Transplantation of cLSC
  Arms: Cultivated Limbal Stem-Cells (cLSC)
Device: Scleral contact lens (SCL) — Scleral contact lens device (SCL) will be used to stabilize and improve ocular surface.
  Arms: Scleral Contact Lens Device (SCL)

SUMMARY:
This phase I study will collect preliminary information on the activity and safety of cLSC. We will investigate the ability to manufacture and transplant cLSC onto the cornea successfully at the time of surgery (feasibility), and have cLSC begin to populate the ocular surface (efficacy) without serious adverse events (safety).

DETAILED DESCRIPTION:
20 patients with severe to total Limbal Stem Cell Deficiency (LSCD) in one eye attributable to injury or ocular surgery. The first 5 eyes will receive the cLSCs to determine the feasibility and safety. Then the subsequent 15 eyes will be randomized into cLSC group and a scleral lens treatment (SCL) control group in a 2:1 ratio in blocks of 3 or 6 using a random number generator.

ELIGIBILITY:
Main inclusion Criteria:

1. Male or female ≥18 years of age.
2. Best corrected visual acuity in the affected eye of 20/160 or less.
3. Documentation of a LSCD diagnosis and the central cornea is affected.
4. Absence of lagophthalmos and eyelid abnormality
5. Adequate forniceal depth is ≥ 5 mm.
6. LSCD fails to resolve by surgical treatments of the ocular surface during the previous 6 months of screening visit.
7. If the etiology of LSCD is due to chemical injury, a minimal interval of 1 year since the initial chemical injury is required.
8. A Schirmer test result at 5 minute of ≥5 mm of wetting.
9. Absence of active infectious keratitis in either eye at the Enrollment Visit.
10. Have a life expectancy ≥ 2 years after enrollment.

Main exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Exposure keratopathy or lagophthalmos of the study eye.
4. Persistent severe ocular surface inflammation and/or meibomian gland dysfunction
5. Chemical injury occurred less than 12 months ago.
6. Presence of ocular surface tumor.
7. Uncontrolled diabetes with last hemoglobin A1C (HgA1C) >8.5.
8. Presence of known allergies to any of the cLSC components.
9. Current participation in another simultaneous medical investigation or trial.
10. Unable to be compliant with or complete the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2027-02-04 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety of cLSC Transplant pertaining to Infection and/or Corneal Perforation | 12 months for all participants
  Safety assessed by incidence of Serious Adverse Events (SAEs) directly related to cLSC: infection and/or corneal perforation.
Feasibility of cLSC Transplant pertaining to Manufacturing meeting Release Criteria | 12 months for all participants
  Feasibility assessed by successful manufacturing of cLSC from biopsy that meets release criteria.
Feasibility of cLSC Transplant pertaining to Manufacturing without Contamination | 12 months for all participants
  Feasibility assessed by successful cLSC manufacturing without contamination.

SECONDARY OUTCOMES:
Changes in the Area of Corneal Epithelial Defect | At 6 months and 12 months in both cLSC and the control groups
  Evaluate changes in the area of corneal epithelial defect (ED) or lack of ED.
Changes in the Clinical Score | At 6 months and 12 months in both cLSC and the control groups
  Evaluate changes in the clinical score determined by slit lamp examination using fluorescein staining and confocal imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Deng, MD, PhD, Principal Investigator — Stein Eye Institute UCLA
Locations (1):
- University of California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No